CLINICAL TRIAL: NCT05059496
Title: Effects of Hamstring Stretching Using Pressure Biofeedback Unit in Patients With Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00854 Maryum Rahim
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain
Keywords: Hamstring length; Low back Pain; Pressure Biofeedback unit
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hamstring stretching with Pressure Biofeedback Unit (Experimental): Hot pack, Hamstring stretching with Biofeedback unit, TENS
  Interventions: Other: Hamstring stretching with Pressure Biofeedback Unit
- Hamstring stretching with out Pressure Biofeedback Unit (Active Comparator): Hot pack, Hamstring stretching without Biofeedback unit, TENS
  Interventions: Other: Hamstring stretching with out Pressure Biofeedback Unit

INTERVENTIONS:
Other: Hamstring stretching with Pressure Biofeedback Unit — Hot Pack 15 mins/1 set/ (3 days/week), Hamstring stretching with Pressure Biofeedback Unit 30 secs hold/ 15 secs rest/ 3 sets/ (3 days/week), TENS 15 mins/ 1 set/ (3 days/week). A total of 4 weeks (12 sessions, 3 days/ week) were given each consisting of 35 mins.
  Arms: Hamstring stretching with Pressure Biofeedback Unit
Other: Hamstring stretching with out Pressure Biofeedback Unit — Hot Pack 15 mins/1 set/ (3 days/week), Hamstring stretching without Pressure Biofeedback Unit 30 secs hold/ 15 secs rest/ 3 sets/ (3 days/week), TENS 15 mins/ 1 set/ (3 days/week). A total of 4 weeks (12 sessions, 3 days/ week) were given each consisting of 35 mins.
  Arms: Hamstring stretching with out Pressure Biofeedback Unit

SUMMARY:
To determine the effects of Hamstring stretching using a pressure Biofeedback unit on muscle length, pain, and functional status in patients with low back pain.

DETAILED DESCRIPTION:
Several studies have been conducted regarding hamstring stretching with the pelvis anteriorly tilted for treating low back pain but there is very little evidence regarding the use of a pressure biofeedback unit for maintaining anterior pelvic tilt so this study aims to find out whether the hamstring stretching while maintaining anterior pelvic tilt using pressure biofeedback is more effective than hamstring stretching without using pressure biofeedback in patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific low back pain
* Chronic pain > 3 months
* Participants having (ODI) score minimum 20% to 40%
* Participants with hamstrings shorter than 70 degrees bilaterally
* Participants who scored 3 or more than 3 on the Numeric Pain Rating Scale (NPRS)

Exclusion Criteria:

* History of fracture and surgery
* Patients with osteoarthritis and spondylolisthesis
* Patients with systemic disease except for diabetes mellitus and hypertension
* Patients with disc herniation and leg length discrepancy
* Pregnant females
* Participants with severe back pain or excessive lumber lordosis

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Hamstring Length | 12 days
  Changes from baseline, Hamstring length was measured through Goniometer. Normal value of Active knee extension is 90 degree with 90 degree hip flexion. Values less than 70 degree knee extension represents hamstring tightness.

SECONDARY OUTCOMES:
Pain through NPRS | 12 days
  Changes from baseline, Pain was measured through Numeric pain rating scale. 0 represents "no pain" and 10 "worst pain possible".
Functional Status | 12 days
  Changes from baseline, Functional status was measured through Oswestry Disability Index. 0-20 shows "minimal disability", 21-40 "moderate disability", 41-60 "severe disability", 61-80 "crippled" and 81-100 "bed bound patients".

CONTACTS AND LOCATIONS:
Overall Officials: Momena Shahzad, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No